CLINICAL TRIAL: NCT06987162
Title: Comparative Effects of Percussive Therapy and Instrument-Assisted Soft Tissue Mobilization On Pain, Muscle Flexibility and Function in Patients With Chronic Non-Specific Low Back Pain.
Brief Title: Percussive Therapy vs Instrument-Assisted Soft Tissue Mobilization on Chronic Non-Specific Low Back Pain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0174 Hamad
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: Low Back Pain,; IASTM; Thera gun; Percussive Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percussive Therapy (Experimental): PT will be performed by the same researcher using a hand-held massage gun, tapping at a frequency of 30 Hz (rotational speed 1800 rpm/min) with a flat massage head. Each percussive massage session will last for 15 minutes. This frequency of 30 Hz is chosen based on its effectiveness for myofascial release and previous studies have indicated that a 15-minute duration of back massage is beneficial
  Interventions: Other: Percussive Therapy
- Instrument-Assisted Soft Tissue Mobilization (Active Comparator): The Graston group performed as IASTM during 4 weeks. After warmup session, Friction free oil or gel was used to facilitate the device to move over the skin. Gua Sha tools were used. The instrument was kept at 45°, moved over the skin from cranial to caudal for 40-120 Sec on the back, while patients were lying in the prone position.The mobilization with sweeping strokes followed by fanning strokes were applied over the Erector spinae, quadratus lumborum, scrolling the device on the muscle belly from the posterior fascia and sacrum.
  Interventions: Other: Instrument-Assisted Soft Tissue Mobilization

INTERVENTIONS:
Other: Percussive Therapy — PT will be performed by the same researcher using a hand-held massage gun, tapping at a frequency of 30 Hz (rotational speed 1800 rpm/min) with a flat massage head. Each percussive massage session will last for 15 minutes. This frequency of 30 Hz is chosen based on its effectiveness for myofascial release and previous studies have indicated that a 15-minute duration of back massage is beneficial
  Arms: Percussive Therapy
Other: Instrument-Assisted Soft Tissue Mobilization — The Graston group performed as IASTM during 4 weeks. After warmup session, Friction free oil or gel was used to facilitate the device to move over the skin. Gua Sha tools were used. The instrument was kept at 45°, moved over the skin from cranial to caudal for 40-120 Sec on the back, while patients were lying in the prone position.The mobilization with sweeping strokes followed by fanning strokes were applied over the Erector spinae, quadratus lumborum, scrolling the device on the muscle belly from the posterior fascia and sacrum.
  Arms: Instrument-Assisted Soft Tissue Mobilization

SUMMARY:
This study compares percussive therapy and instrument-assisted soft tissue mobilization (IASTM) for chronic non-specific low back pain (CNSLBP). Percussive therapy uses handheld devices for rapid pressure pulses to promote muscle relaxation and pain relief. IASTM employs specialized tools to massage tissues, break down scar tissue, and enhance flexibility and blood flow. The research aims to assess their effects on pain reduction, muscle flexibility, and functional improvement in CNSLBP patients.

DETAILED DESCRIPTION:
This study will be a randomized Clinical trial in which 52 sample size will be taken. This randomized clinical trial aims to compare the effects of Percussive Therapy (PT) and Instrument-Assisted Soft Tissue Mobilization (IASTM) on pain, muscle flexibility, and function in patients with chronic non-specific low back pain at Riphah International University, Pakistan. Using a Non probability convenient sampling method, participants aged 18-50 years with chronic non-specific low back pain will be selected based on inclusion and exclusion criteria. In both groups the warm-up sessions included arm circular movements with eight repetitions forward and eight repetitions backward, while standing on the feet the subjects were asked to stand on wide-based feet and move the right and left arm forward in a swing way in a circular motion, and that backward They will be equally divided into two groups using a random number generator table. Group A will receive Percussive Therapy, while Group B will receive Instrument-Assisted Soft Tissue Mobilization. These exercises will continue for 4 weeks, 4 days per week. Outcome measures, including the Numerical Pain Rating Scale (NPRS) for pain intensity, Oswestry Disability Index (ODI) for functional impairment, Sit and Reach Test for back flexibility, will be assessed at baseline and after four weeks of intervention.

Ethical approval will be obtained from the Ethical Committee of Riphah International University, and informed consent will be secured from all participants. The primary outcomes will focus on pain intensity and functional disability, while secondary outcomes will include muscle flexibility and spinal mobility. Data analysis will be performed using SPSS version 25.

The findings are expected to provide valuable insights into the comparative efficacy of these manual therapy techniques, informing clinical practice and improving patient outcomes in the management of chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age Range of 18 To 50 Years.
* Presence of Chronic Low Back Pain for more than 3 months
* Pain level according to Visual Analogue Scale greater or equal to 3

Exclusion Criteria:

* Trauma History: Patients with A History of Trauma Were Excluded
* Diabetic Patients
* Recent History of Trauma
* Any Neurological or Musculoskeletal Disorder of the Upper Limb/Lower Limb Osteoporosis
* Lumbar Compression Fracture
* Spondylolisthesis; Spondylosis; Spinal Deformities; History of Spinal Surgeries

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Sit and Reach test | 4 weeks
  To perform this test, all subjects sat with their heels firmly against the testing box. Subjects kept their knees extended and placed their right hand over the left, with the long fingers even, and reached forward as far as they could by sliding their hands along the measuring board indicated in centimeters how far beyond the toes each individual reached. The score(in centimeters) is the greatest distance contacted by the fingertips past the toes. 3 trials were performed, and the average was used for data analysis.

SECONDARY OUTCOMES:
NPRS | 4 WEEKS
  NPRS:
  The NPRS is frequently employed to measure pain intensity, in which patients are asked to select a number (from 0 to 10) to represent their pain severity.

OTHER OUTCOMES:
Oswestry Disability Index (ODI): | 4 weeks
  The ODI is a ten-item questionnaire that assesses the disabling effects of LBP on activities of daily living (ADL). It is a reliable and valid self-reported questionnaire that lasts 5 min for the patient to complete the measure and a few minutes for the examiner to calculate the scores.
  Each item is scored from 0 to 5, and the summation of the ten scores is stated as a percentage of the maximum score; therefore, it ranges from 0 (no disability) to 100 (maximum disability)

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Phd Scholar, Principal Investigator — Riphah International University
Locations (1):
- Zafar Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agnus Tom A, Rajkumar E, John R, Joshua George A. Determinants of quality of life in individuals with chronic low back pain: a systematic review. Health Psychol Behav Med. 2022 Jan 5;10(1):124-144. doi: 10.1080/21642850.2021.2022487. eCollection 2022. PMID 35003902
- [Background] Peck J, Urits I, Peoples S, Foster L, Malla A, Berger AA, Cornett EM, Kassem H, Herman J, Kaye AD, Viswanath O. A Comprehensive Review of Over the Counter Treatment for Chronic Low Back Pain. Pain Ther. 2021 Jun;10(1):69-80. doi: 10.1007/s40122-020-00209-w. Epub 2020 Nov 4. PMID 33150555
- [Background] Du S, Liu W, Cai S, Hu Y, Dong J. The efficacy of e-health in the self-management of chronic low back pain: A meta analysis. Int J Nurs Stud. 2020 Jun;106:103507. doi: 10.1016/j.ijnurstu.2019.103507. Epub 2019 Dec 24. PMID 32320936
- [Background] Frizziero A, Pellizzon G, Vittadini F, Bigliardi D, Costantino C. Efficacy of Core Stability in Non-Specific Chronic Low Back Pain. J Funct Morphol Kinesiol. 2021 Apr 22;6(2):37. doi: 10.3390/jfmk6020037. PMID 33922389
- [Background] Patel R, Patel AJJADMS. Effect of Theragun on the improvement of back flexibility: A case study. 2020;19(5):15-6.
- [Background] Mansuri U, Patel SJIJSR. Effectiveness of Theragun and ergonomic advice in patients with low back pain among bus drivers-A randomized controlled trial. 2021;10(4):50-3.
- [Background] Jain P, Saharan AK, Vishnoi CS, Bhati MPS, Sharma PJGAR, Reviews. Single IASTM and cupping therapy session improves pain and disability in patients with non-specific low back pain. 2022;11(3):045-50.
- [Background] Johnson S. The Effects of Instrument Assisted Soft Tissue Mobilization: A Systematic Review and Meta-Analysis. 2023.
- [Background] Grase M, Elhafez HM, Abdellatif MM, Genedi AF, Mahmoud MAJPQ. Effect of instrument assisted soft tissue mobilization versus kinesiotape for chronic mechanical low back pain: a randomized controlled trial. 2023;31(2):27-33.
- [Background] Çakmak Ö, Atıcı E, Gülşen MJTFvRD. The effects of instrument-assisted soft tissue mobilization and kinesio taping on pain, functional disability and depression in patients with chronic low back pain: a randomized trial. 2022;33(3):179-86.